CLINICAL TRIAL: NCT00412867
Title: Post-marketing Clinical Study of Alteplase for Acute Ischemic Stroke (Phase 4)
Brief Title: Post-marketing Clinical Study of Alteplase for Acute Ischemic Stroke （Japan Alteplase Clinical Trial Ⅱ：J-ACT Ⅱ）
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 527-0611; NCT00412945 (obsolete NCT alias)
Record Dates: First submitted 2006-12-17; First posted 2006-12-19 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Cerebral Infarction; acute ischemic stroke; Brain ischemia
MeSH Terms: conditions — Stroke; Cerebral Infarction; Ischemic Stroke; Brain Ischemia | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alteplase (Experimental): 0.6mg/kg intravenous alteplase with 10% being administered as a bolus followed by continuous infusion of the remainder over 1 hour
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — 0.6 mg/kg of Alteplase is intravenously administered
  Other Names: Tissue Plasminogen Activator; GRTPA; ACTIVACIN

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of intravenously administered alteplase in patients with acute ischemic stroke based on the rate of recanalization assessed by magnetic resonance angiography (MRA), the rate of patients with a modified Rankin Scale (mRS) score of 0-1, and the incidence of symptomatic intracranial hemorrhage (sICH), in comparison with the data reported in the current literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke within 3 hours of onset, with a clearly defined time of onset.
* Patients who have been revealed to have occlusion on one side of the middle cerebral artery (M1 or M2 portion) on MRA before the start of treatment.
* Patients for whom consent has been obtained from either themselves or from their legally acceptable representatives in written form.

Exclusion Criteria:

* Patients with very light neurological symptoms (an NIHSS score of <= 4) or with rapidly improving symptoms before the start of treatment.
* Patients with serious neurological disorders (an NIHSS score of >= 23), or serious consciousness disorders (a Japan Coma Scale score of >= 100) before the start of treatment.
* Patients with functional disorders (a mRS score of >= 2) before stroke onset.
* Patients who have been administered drugs that are not allowed to be administered concomitantly with alteplase (other thrombolytic agents) after the stroke onset.
* Patients who have been revealed to have extensive early ischemic change (an Alberta Stroke Program Early CT score of <= 6) on computed tomography (CT) before treatment.
* Patients who have been revealed to have obvious occlusion in the blood vessel except for the middle cerebral artery on MRA before treatment.
* Patients who are forbidden to undergo magnetic resonance imaging (MRI).
* Patients who are defined as having cerebral hemorrhage or subarachnoid hemorrhage (SAH) on CT before treatment.
* Patients whose symptoms suggest SAH.
* Patients with hemorrhage (gastrointestinal hemorrhage, urinary hemorrhage, retroperitoneal hemorrhage, or hemoptysis).
* Patients with a platelet count below 100,000/mm3.
* Patients with fasting blood glucose levels of < 50 mg/dL or > 400 mg/dL.
* Patients whose activated partial thromboplastin time (APTT) is prolonged due to heparin administration within 48 hours before stroke onset.
* Patients who have been administered oral anticoagulants with values of the international normalized ratio of prothrombin time (PT-INR) of > 1.7.
* Patients who have a systolic blood pressure of > 185 mmHg or a diastolic blood pressure of > 110 mmHg.
* Patients who need antihypertensive therapy (e.g. continuous infusion of antihypertensive drug etc.) to lower blood pressure below those limits under the preceding article.
* Patients who have a history of intracranial hemorrhage, or who have a disease considered to increase the risk of intracranial hemorrhage such as an intracranial tumor, cerebral aneurysm, or intracranial arteriovenous malformation, etc.
* Patients who have a history of stroke within 3 months before onset.
* Patients who were operated on or injured their head or spinal cord within 3 months before onset.
* Patients who have a history of gastrointestinal or urinary tract hemorrhage within 21 days before onset.
* Patients who had a major surgery or serious trauma (except for head or spinal cord trauma) within 14 days before onset.
* Patients who have a history of organ biopsy, arterial puncture, or lumbar puncture within 10 days before onset.
* Patients with severe hepatic dysfunction or severe renal dysfunction.
* Patients with acute pancreatitis.
* Patients who had a seizure at the onset of stroke.
* Patients who have a history of hypersensitivity to protein preparations.
* Patients who are lactating, pregnant, probably pregnant, or menstruating.
* Patients with malignant tumors.
* Patients with acute myocardial infarction (AMI) or pericarditis after AMI.
* Patients with concurrent infectious endocarditis, moyamoya disease (Willis circle occlusion syndrome), aortic dissection, or neck trauma, etc.
* Patients with strong suspicion of ischemic cerebrovascular disorder caused by non-thrombotic occlusion or any other hemodynamic condition.
* Patients judged to be difficult in monitoring for 3 months by their physician.
* Patients who have participated in other clinical trials during the last 3 months.
* In addition to the above exclusion criteria, patients judged to be inadequate to participate in this study by their physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takenori Yamaguchi, M.D., Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- Investigational site 01, Hokkaido, Japan

REFERENCES:
- [Result] Mori E, Minematsu K, Nakagawara J, Yamaguchi T, Sasaki M, Hirano T; Japan Alteplase Clinical Trial II Group. Effects of 0.6 mg/kg intravenous alteplase on vascular and clinical outcomes in middle cerebral artery occlusion: Japan Alteplase Clinical Trial II (J-ACT II). Stroke. 2010 Mar;41(3):461-5. doi: 10.1161/STROKEAHA.109.573477. Epub 2010 Jan 14. PMID 20075341
- [Derived] Hirano T, Sasaki M, Mori E, Minematsu K, Nakagawara J, Yamaguchi T; Japan Alteplase Clinical Trial II Group. Residual vessel length on magnetic resonance angiography identifies poor responders to alteplase in acute middle cerebral artery occlusion patients: exploratory analysis of the Japan Alteplase Clinical Trial II. Stroke. 2010 Dec;41(12):2828-33. doi: 10.1161/STROKEAHA.110.594333. Epub 2010 Oct 28. PMID 21030700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alteplase
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alteplase
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Valid Recanalization Assessed by Magnetic Resonance Angiography (MRA)
Description: Recanalization was evaluated according to the modified Mori grade: Grade 0, no reperfusion; Grade 1, movement of thrombus not associated with any flow improvement; Grade 2, partial (branch) recanalization in <50% of the branches in the occluded-arterial territory; Grade 3, nearly complete recanalization with reperfusion in ≥50% of the branches in the occluded-arterial territory.
  The recanalization rate was estimated by regarding Grades 2 and 3 as valid recanalization.
Time Frame: within 6 hours, from 24 to 36 hours after onset
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 58
participants
  within 6 hours after onset | 30
  from 24 to 36 hours after onset | 40

2. Primary Outcome: Number of Patients With a Modified Rankin Scale (mRS) Score of 0-1 a 3 Months
Description: The number of patients with an mRS score of 0-1. The mRS has 6 items, where 0 = No symptoms at all, 1 = No significant disability despite symptoms, 2 = Slight disability, 3 = Moderate disability, 4 = Moderately severe disability, 5 = Severe disability. The higher scores reflect increased disability.
Time Frame: 3 months after onset
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 58
participants | 27

3. Primary Outcome: Number of Patients With Symptomatic Intracranial Hemorrhage (sICH) Within 36 Hours
Description: The number of patients with sICH
Time Frame: within 36 hours after starting treatment
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 58
participants | 0

4. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS) Score
Description: from 0 (normal) to 40 (most severe)
Time Frame: within 6 hours, from 24 to 36 hours, 3 months after onset.
Population: Two participants (from 24 to 36 hours) and four participants (3 months after onset) were excluded from analysis because of dropouts or missing data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Alteplase
Number analyzed (Participants) | 58
units on a scale
  within 6 hours | 8.5 [0 to 20]
  from 24 to 36 hours: number analyzed (Participants) | 56
  from 24 to 36 hours | 7.0 [0 to 22]
  3 months after onset: number analyzed (Participants) | 54
  3 months after onset | 1.5 [0 to 32]

5. Secondary Outcome: Barthel Index (BI)
Description: from 100 (Independent) to 0 (full assistance)
Time Frame: the day of discharge within 3 months after onset, and 3 months after onset
Population: Eleven participants (the day of discharge within 3 months after onset) and four participants (3 months after onset) were excluded from analysis because of dropouts or missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alteplase
Number analyzed (Participants) | 58
units on a scale
  the day of discharge within 3 months after onset: number analyzed (Participants) | 47
  the day of discharge within 3 months after onset | 76.2 (32.4)
  3 months after onset: number analyzed (Participants) | 54
  3 months after onset | 77.8 (33.2)

6. Secondary Outcome: Percentage of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: 3 months
Measure: Number; unit: percentage of patients
Arm/Group | Alteplase
Number analyzed (Participants) | 58
percentage of patients
  Percentage of Patients with Adverse Events | 96.6
  Percentage of Patients with Adverse Drug Reactions | 41.4

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Alteplase (Non-Haemorrhage); Alteplase (Haemorrhage): 0.6mg/kg intravenous alteplase with 10% being administered as a bolus followed by continuous infusion of the remainder over 1 hour
Arm/Group | Alteplase (Non-Haemorrhage) | Alteplase (Haemorrhage)
Serious Adverse Events (participants affected / at risk) | 12/58 | 1/58
Other Adverse Events (participants affected / at risk) | 51/58 | 25/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase (Non-Haemorrhage) (N=58) | Alteplase (Haemorrhage) (N=58)
Cardiac failure (Cardiac disorders) | 2 | 0
Sick sinus syndrome (Cardiac disorders) | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 4 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase (Non-Haemorrhage) (N=58) | Alteplase (Haemorrhage) (N=58)
Atrial fibrillation (Cardiac disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Tricuspid valve incompetence (Cardiac disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 27 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0
Pyrexia (General disorders) | 5 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 10 | 0
Liver disorder (Hepatobiliary disorders) | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0
Urinary tract infections (Infections and infestations) | 10 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 0
Blood fibrinogen increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 3 | 0
Blood urine present (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 2 | 0
Protein urine present (Investigations) | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 21
Headache (Nervous system disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 13 | 0
Restlessness (Psychiatric disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Neurogenic bladder (Renal and urinary disorders) | 6 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor's consent must be obtained in advance if the investigator or other study-related personnel in the study center intend to publish information obtained via this study at a scientific conference or similar venue.